CLINICAL TRIAL: NCT04511572
Title: Improving the Outcome of Chronic Subdural Hematoma by Embolization of Middle Meningeal Artery (ELIMINATE)
Brief Title: Embolization of Middle Meningeal Artery in Chronic Subdural Hematoma
Acronym: ELIMINATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. W.Peter Vandertop, chair Neurosurgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC Eliminate
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Subdural Hematomas
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care: burr hole surgery (No Intervention): Patients who have had burr hole evacuation for symptomatic chronic subdural hematomas will be followed in the outpatient clinic after hospital discharge at 8, 16 and 24 weeks with a follow-up CT-scan of the head in addition to assessment of mRS, MOCA, mNIHSS, Markwalder score, SF-36, EQ-5D-5L, ALDS, iMCQ and iPCQ.
- embolisation middle meningeal artery (Active Comparator): Besides standard treatment those patient who are allotted to the intervention group will receive embolization of the middle meningeal artery until 72 hours after burr hole evacuation. After hospital discharge follow-up is at 8, 16 and 24 weeks with a follow-up CT-scan of the head in addition to assessment of mRS, MOCA, mNIHSS, Markwalder score, SF-36, EQ-5D-5L, ALDS, iMCQ and iPCQ.
  Interventions: Procedure: embolization of the middle meningeal artery

INTERVENTIONS:
Procedure: embolization of the middle meningeal artery — The embolization procedure will be as follows: first femoral artery access will be obtained by using a 5 French micropuncture kit and common carotid and external carotid angiography is performed using a standard 5 French diagnostic catheter. A microcatheter is then advanced selectively under roadmap guidance into the middle meningeal artery (MMA), and MMA angiography is performed to evaluate for potential dangerous anastomoses such as the orbital branch to the ophthalmic artery. Embolization is performed using polyvinyl alcohol particles (100 microns in diameter) under blank fluoroscopic roadmap while carefully avoiding reflux. Particles are infused until lack of anterograde flow into the MMA branches is demonstrated on angiography, and the catheters are removed [31]. The procedure is performed under local anesthesia.
  Arms: embolisation middle meningeal artery

SUMMARY:
Chronic subdural hematoma (cSDH) is a common neurological affliction which affects mostly frail and elderly patients. Surgical evacuation by using burr hole craniostomy (BHC) is the most frequently used treatment but carries a recurrence rate varying between 10-30% in the literature. Especially in this frail population re-operation is undesirable. Embolization of the middle meningeal artery is an adjuvant treatment which has been reported in multiple case reports and larger case series, showing a beneficial effect on recurrence rate, reducing it to <5%, without complications.

Objectives: Primary: To evaluate whether additional embolization of the middle meningeal artery after surgery for cSDH reduces the recurrent surgery rate. Secondary: to evaluate whether the use of middle meningeal artery embolization after surgical treatment in symptomatic cSDH patients increases quality of life (SF-36 and the EQ-5D-5L), performance in activities of daily living (AMC Linear Disability Score), functional outcome (mRS), cognitive functioning (MOCA) and reduces mortality, occurrence of complications, recurrence rate, size and volume of the hematoma, neurological impairment (mNIHSS, Markwalder score) and the use of care and health-related costs (iMCQ and iPCQ).

Study design: Multicenter, randomized controlled open-label superiority trial. Study population: Patients diagnosed with a cSDH who require surgery. Intervention: The intervention group will receive embolization in addition to standard surgical treatment. The control group will receive surgery only.

Main study endpoint: The number of patients who require reoperation within 24 weeks after the intervention.

Symptomatic cSDH patients will undergo peri-operative embolization of the middle meningeal artery until 72 hours after surgical treatment. Complications are monitored during hospital admission and follow-up. Radiological and clinical follow-up is at eight, 16 and 24 weeks post-intervention with a CT-scan of the head and assessment of mRS, MOCA, mNIHSS, Markwalder score, SF-36, EQ-5D-5L, ALDS, iMCQ and iPCQ. Standard care after surgery entails outpatient follow-up with on average two CT-scans, indicated by clinical signs and symptoms.

DETAILED DESCRIPTION:
Chronic subdural hematoma A chronic subdural hematoma (cSDH) is a bleeding of the bridging veins between the dura mater and the arachnoid.

Subdural hematomas are one of the most common forms of hemorrhage affecting mostly elderly people. The estimated incidence in Western countries is 8.1 per 100,000 per year in patients aged 65 years or older, but increases to 58/100,000/year for those aged 70 years or older. With the elderly population growing, the incidence of cSDH is expected to double by 2030. CSDH presents itself as an heterogeneous disease with various symptoms. Most common are gait disturbances, focal deficits, headaches and hemiparesis. Risk factors for occurrence are chronic alcoholism, male gender and anticoagulation and antiplatelet therapy. CSDH is a challenging disease of which the pathophysiology is not completely clear. Even though cSDH initially arises due to tearing of the bridging veins, its chronicity likely has an arterial origin. At first a subdural hematoma forms after a (minor) head trauma. The hematoma persists due to failure of the reparative and absorbing mechanisms. The current hypothesis states that the inability of the human body to heal the hematoma is due to increased neovascularization in the subdural membrane of the hematoma. This leads to repeated micro hemorrhages and further increase in fibrinolytic activity, which makes the body unable to stop recurrent microbleeds. Repeated micro hemorrhages are caused by collateral blood vessels originating from the middle meningeal artery. The correlation between the cycle of re-bleeding and fibrinolysis, and reabsorption of the subdural collection will determine whether the cSDH will resolve, persist or enlarge.

Treatment options The first treatment option for mildly symptomatic cSDH is a conservative 'wait-and-scan' approach in which the patient is followed with CT-scans and outpatient clinic visits. The majority (75%) of these conservatively managed patients however, eventually still require surgery (own data). Medical treatment is a second non-surgical treatment option currently being studied in large RCTs, for instance with steroids (dexamethasone), mannitol, tranexamic acid (TORCH-study), statins and ACE-inhibitors.

Surgical treatment is most frequently used in symptomatic patients with a cSDH as surgery provides instant decompression of the brain and rapid relief of (life-threatening) symptoms. However, surgery is costly and in these often frail patients with multi-morbidity, surgery comes with significant risks for future cognitive functioning and therefore loss of independence. Furthermore, recurrence rates after surgery range from 9-30%, resulting in frequent re-operations. Therefore, the optimal treatment for cSDH remains a 'burning clinical question' for which neurologists and neurosurgeons do not have evidence-based answers. Multiple studies have described successful treatment with embolization of the middle meningeal artery as an adjunct to surgical evacuation. The goal of embolization is to devascularize the subdural membranes to a sufficient extent such that the balance is shifted from the continued rebleeding and accumulation of blood products towards reabsorption of the subdural effusion. The use of embolization in cSDH patients was first reported in 2000, and since then multiple case reports, case series and cohort studies have been published investigating the safety and effectiveness. The largest cohort study compared 72 patients with embolization (as sole treatment or with surgical treatment combined) to 469 (retrospectively) non-surgical treated patients. In this study no complications were reported and only one patient needed repeat surgery. A relatively large case series of 60 patients was reported, again with no complications and a success rate of 92% (patients who were able to avoid surgery). Recent systematic reviews on middle meningeal artery embolization highlight the lower recurrence and complication rate in all embolization cases (<5% and 0%, respectively). Nevertheless, these results are based on non-randomized studies with moderate quality and a small sample size. The effect of embolization as an adjunct to surgical evacuation has never been evaluated in a randomized controlled trial.

In conclusion, although surgery is still the primary treatment option for the majority of patients with cSDH, it carries a significant risk of additional morbidity and mortality and has a relatively high risk of treatment failure. In the aging population, comorbidities are more frequent and the risk of peri-operative complications is acknowledged, limiting a favorable clinical outcome. Middle meningeal artery embolization appears to be a promising adjunct therapy to surgery, which might reduce the necessity for repeat surgical treatment and improve clinical outcome is this vulnerable patient group.

ELIGIBILITY:
Inclusion Criteria:

* · CT-confirmed diagnosis of chronic Subdural Hematoma;

  * Primary surgical treatment based on clinical symptoms (progressive neurological deficits).

Exclusion Criteria:

* · Significant contraindication to angiography (eg. allergy for contrast);

  * Structural causes for subdural hemorrhage, e.g. arachnoid cysts, cortical vascular malformations and a history of cranial surgery in the previous 365 days;
  * Inability to obtain informed consent from the patient or legal representative (when the patient has a depressed level of consciousness), including language barrier;
  * Monocular blindness on contralateral side of the hematoma;

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Reoperation | 8 weeks after discharge.
  Number of patients who require a reoperation for recurrent cSDH
Reoperation | 16 weeks after discharge.
  Number of patients who require a reoperation for recurrent cSDH
Reoperation | 24 weeks after discharge.
  Number of patients who require a reoperation for recurrent cSDH

SECONDARY OUTCOMES:
Hematoma volume reduction | 8 weeks after discharge.
  hematoma volumes are measured on CT-scan of the head and compared to pre-operative volume
Hematoma volume reduction | 16 weeks after discharge.
  hematoma volumes are measured on CT-scan of the head and compared to pre-operative volume
Hematoma volume reduction | 24 weeks after discharge.
  hematoma volumes are measured on CT-scan of the head and compared to pre-operative volume
Complications | 8 weeks after discharge.
  Number of complications will be monitored
Complications | 16 weeks after discharge.
  Number of complications will be monitored
Complications | 24 weeks after discharge.
  Number of complications will be monitored
modified National Institute Health Stroke Scale score | 8 weeks after discharge.
  Neurological impairment measurement using mNIHSS; score 0 (no symptoms) to 31 (severe stroke)
modified National Institute Health Stroke Scale score | 16 weeks after discharge.
  Neurological impairment measurement using mNIHSS; score 0 (no symptoms) to 31 (severe stroke)
modified Rankin Scale score | 24 weeks after discharge.
  functional outcome measurement using mRS; score 0 (no symptoms) to 5 (severe handicap)
modified National Institute Health Stroke Scale score | 24 weeks after discharge.
  Neurological impairment measurement using mNIHSS; score 0 (no symptoms) to 31 (severe stroke)
Montreal Cognitive Assessment | 8 weeks after discharge.
  cognitive functioning measurement using MOCA; score 0 (severe deficit to 30 (no deficit)
Montreal Cognitive Assessment | 16 weeks after discharge.
  cognitive functioning measurement using MOCA; score 0 (severe deficit to 30 (no deficit)
Montreal Cognitive Assessment | 24 weeks after discharge.
  cognitive functioning measurement using MOCA; score 0 (severe deficit to 30 (no deficit)
mortality | 8 weeks after discharge.
  mortality rate
mortality | 16 weeks after discharge.
  mortality rate
mortality | 246 weeks after discharge.
  mortality rate
Activities of Daily Living Scale | at 24 weeks after discharge.
  Assesses functional independence, generally in stroke patients; score 0 (totally dependent to 100 (completely independent)
Short Form Health Survey | at 24 weeks after discharge.
  Quality of life measurement using a 36-item, patient-reported survey of patient health; consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
EuroQol (EQ-5D-5L) questionnaire | at 24 weeks after discharge.
  Quality of life measurement:The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Medical Consumption questionnaire | at 24 weeks after discharge.
  Care- and health-related costs measurement using a generic instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers and can be complemented with extra questions that are relevant for specific study populations.
Productivity Cost Questionnaire | at 24 weeks after discharge.
  Care- and health-related costs measurement using a generic instrument for measuring medical costs
Markwalder grading scale score | at eight weeks after discharge
  Neurological impairment measurement using the Markwalder grading scale; score 0 (neurologically normal) to 4 (Comatose with absent motor responses to painful stimuli, decerebrate or decorticate posturing)
Markwalder grading scale score | at 16 weeks after discharge
  Neurological impairment measurement using the Markwalder grading scale; score 0 (neurologically normal) to 4 (Comatose with absent motor responses to painful stimuli, decerebrate or decorticate posturing)
Markwalder grading scale score | at 24 weeks after discharge
  Neurological impairment measurement using the Markwalder grading scale; score 0 (neurologically normal) to 4 (Comatose with absent motor responses to painful stimuli, decerebrate or decorticate posturing)

CONTACTS AND LOCATIONS:
Overall Officials: William P. Vandertop, MD PhD, Study Chair — Amsterdam Universities Medical Centers
Locations (1):
- Amsterdam university medical Centers, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miah IP, Holl DC, Peul WC, Walchenbach R, Kruyt N, de Laat K, Koot RW, Volovici V, Dirven CMF, van Kooten F, Kho KH, den Hertog HM, van der Naalt J, Jacobs B, Groen RJM, Lingsma HF, Dammers R, Jellema K, van der Gaag NA; Dutch Subdural Hematoma Research Group (DSHR). Dexamethasone therapy versus surgery for chronic subdural haematoma (DECSA trial): study protocol for a randomised controlled trial. Trials. 2018 Oct 20;19(1):575. doi: 10.1186/s13063-018-2945-4. PMID 30342554
- [Background] Santarius T, Kirkpatrick PJ, Kolias AG, Hutchinson PJ. Working toward rational and evidence-based treatment of chronic subdural hematoma. Clin Neurosurg. 2010;57:112-22. PMID 21280503
- [Background] Sahyouni R, Goshtasbi K, Mahmoodi A, Tran DK, Chen JW. Chronic Subdural Hematoma: A Historical and Clinical Perspective. World Neurosurg. 2017 Dec;108:948-953. doi: 10.1016/j.wneu.2017.09.064. Epub 2017 Sep 19. PMID 28935548
- [Background] Yang W, Huang J. Chronic Subdural Hematoma: Epidemiology and Natural History. Neurosurg Clin N Am. 2017 Apr;28(2):205-210. doi: 10.1016/j.nec.2016.11.002. Epub 2017 Feb 1. PMID 28325454
- [Background] Holl DC, Volovici V, Dirven CMF, Peul WC, van Kooten F, Jellema K, van der Gaag NA, Miah IP, Kho KH, den Hertog HM, Lingsma HF, Dammers R; Dutch Chronic Subdural Hematoma Research Group (DSHR). Pathophysiology and Nonsurgical Treatment of Chronic Subdural Hematoma: From Past to Present to Future. World Neurosurg. 2018 Aug;116:402-411.e2. doi: 10.1016/j.wneu.2018.05.037. Epub 2018 May 14. PMID 29772364
- [Background] Edlmann E, Giorgi-Coll S, Whitfield PC, Carpenter KLH, Hutchinson PJ. Pathophysiology of chronic subdural haematoma: inflammation, angiogenesis and implications for pharmacotherapy. J Neuroinflammation. 2017 May 30;14(1):108. doi: 10.1186/s12974-017-0881-y. PMID 28558815
- [Background] Waqas M, Vakhari K, Weimer PV, Hashmi E, Davies JM, Siddiqui AH. Safety and Effectiveness of Embolization for Chronic Subdural Hematoma: Systematic Review and Case Series. World Neurosurg. 2019 Jun;126:228-236. doi: 10.1016/j.wneu.2019.02.208. Epub 2019 Mar 13. PMID 30878752
- [Background] Srivatsan A, Mohanty A, Nascimento FA, Hafeez MU, Srinivasan VM, Thomas A, Chen SR, Johnson JN, Kan P. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma: Meta-Analysis and Systematic Review. World Neurosurg. 2019 Feb;122:613-619. doi: 10.1016/j.wneu.2018.11.167. Epub 2018 Nov 24. PMID 30481628
- [Background] Court J, Touchette CJ, Iorio-Morin C, Westwick HJ, Belzile F, Effendi K. Embolization of the Middle meningeal artery in chronic subdural hematoma - A systematic review. Clin Neurol Neurosurg. 2019 Nov;186:105464. doi: 10.1016/j.clineuro.2019.105464. Epub 2019 Aug 10. PMID 31600604
- [Background] Sun TF, Boet R, Poon WS. Non-surgical primary treatment of chronic subdural haematoma: Preliminary results of using dexamethasone. Br J Neurosurg. 2005 Aug;19(4):327-33. doi: 10.1080/02688690500305332. PMID 16455539
- [Background] Soleman J, Nocera F, Mariani L. The conservative and pharmacological management of chronic subdural haematoma. Swiss Med Wkly. 2017 Jan 17;147:w14398. doi: 10.57187/smw.2017.14398. eCollection 2017. PMID 28102879
- [Background] Pang CH, Lee SE, Kim CH, Kim JE, Kang HS, Park CK, Paek SH, Kim CH, Jahng TA, Kim JW, Kim YH, Kim DG, Chung CK, Jung HW, Yoo H. Acute intracranial bleeding and recurrence after bur hole craniostomy for chronic subdural hematoma. J Neurosurg. 2015 Jul;123(1):65-74. doi: 10.3171/2014.12.JNS141189. Epub 2015 Feb 13. PMID 25679282
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Oct;127(4):732-739. doi: 10.3171/2016.8.JNS16134. Epub 2016 Nov 11. PMID 27834599
- [Background] Ducruet AF, Grobelny BT, Zacharia BE, Hickman ZL, DeRosa PL, Andersen KN, Sussman E, Carpenter A, Connolly ES Jr. The surgical management of chronic subdural hematoma. Neurosurg Rev. 2012 Apr;35(2):155-69; discussion 169. doi: 10.1007/s10143-011-0349-y. Epub 2011 Sep 10. PMID 21909694
- [Background] Ban SP, Hwang G, Byoun HS, Kim T, Lee SU, Bang JS, Han JH, Kim CY, Kwon OK, Oh CW. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma. Radiology. 2018 Mar;286(3):992-999. doi: 10.1148/radiol.2017170053. Epub 2017 Oct 10. PMID 29019449
- [Background] Okuma Y, Hirotsune N, Sato Y, Tanabe T, Muraoka K, Nishino S. Midterm Follow-Up of Patients with Middle Meningeal Artery Embolization in Intractable Chronic Subdural Hematoma. World Neurosurg. 2019 Jun;126:e671-e678. doi: 10.1016/j.wneu.2019.02.121. Epub 2019 Mar 4. PMID 30844521
- [Background] Nakagawa I, Park HS, Kotsugi M, Wada T, Takeshima Y, Matsuda R, Nishimura F, Yamada S, Motoyama Y, Park YS, Kichikawa K, Nakase H. Enhanced Hematoma Membrane on DynaCT Images During Middle Meningeal Artery Embolization for Persistently Recurrent Chronic Subdural Hematoma. World Neurosurg. 2019 Jun;126:e473-e479. doi: 10.1016/j.wneu.2019.02.074. Epub 2019 Feb 28. PMID 30825631
- [Background] Link TW, Boddu S, Paine SM, Kamel H, Knopman J. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma: A Series of 60 Cases. Neurosurgery. 2019 Dec 1;85(6):801-807. doi: 10.1093/neuros/nyy521. PMID 30418606
- [Background] Fiorella D, Arthur AS. Middle meningeal artery embolization for the management of chronic subdural hematoma. J Neurointerv Surg. 2019 Sep;11(9):912-915. doi: 10.1136/neurintsurg-2019-014730. Epub 2019 Feb 23. PMID 30798265
- [Background] Mandai S, Sakurai M, Matsumoto Y. Middle meningeal artery embolization for refractory chronic subdural hematoma. Case report. J Neurosurg. 2000 Oct;93(4):686-8. doi: 10.3171/jns.2000.93.4.0686. PMID 11014549
- [Background] Yamamoto S, Asahi T, Akioka N, Kashiwazaki D, Kuwayama N, Kuroda S. Chronic subdural hematoma infected by propionibacterium acnes: a case report. Case Rep Neurol. 2015 Jan 24;7(1):6-14. doi: 10.1159/000371841. eCollection 2015 Jan-Apr. PMID 25759659
- [Background] Tsukamoto Y, Oishi M, Shinbo J, Fujii Y. Transarterial embolisation for refractory bilateral chronic subdural hematomas in a case with dentatorubral-pallidoluysian atrophy. Acta Neurochir (Wien). 2011 May;153(5):1145-7. doi: 10.1007/s00701-010-0891-3. Epub 2010 Dec 2. No abstract available. PMID 21125409
- [Background] Tempaku A, Yamauchi S, Ikeda H, Tsubota N, Furukawa H, Maeda D, Kondo K, Nishio A. Usefulness of interventional embolization of the middle meningeal artery for recurrent chronic subdural hematoma: Five cases and a review of the literature. Interv Neuroradiol. 2015 Jun;21(3):366-71. doi: 10.1177/1591019915583224. Epub 2015 May 26. PMID 26015518
- [Background] Mino M, Nishimura S, Hori E, Kohama M, Yonezawa S, Midorikawa H, Kaimori M, Tanaka T, Nishijima M. Efficacy of middle meningeal artery embolization in the treatment of refractory chronic subdural hematoma. Surg Neurol Int. 2010 Dec 13;1:78. doi: 10.4103/2152-7806.73801. PMID 21206540
- [Background] Matsumoto H, Hanayama H, Okada T, Sakurai Y, Minami H, Masuda A, Tominaga S, Miyaji K, Yamaura I, Yoshida Y. Which surgical procedure is effective for refractory chronic subdural hematoma? Analysis of our surgical procedures and literature review. J Clin Neurosci. 2018 Mar;49:40-47. doi: 10.1016/j.jocn.2017.11.009. Epub 2017 Dec 20. PMID 29274740
- [Background] Link TW, Schwarz JT, Paine SM, Kamel H, Knopman J. Middle Meningeal Artery Embolization for Recurrent Chronic Subdural Hematoma: A Case Series. World Neurosurg. 2018 Oct;118:e570-e574. doi: 10.1016/j.wneu.2018.06.241. Epub 2018 Jul 6. PMID 30257310
- [Background] Kim E. Embolization Therapy for Refractory Hemorrhage in Patients with Chronic Subdural Hematomas. World Neurosurg. 2017 May;101:520-527. doi: 10.1016/j.wneu.2017.02.070. Epub 2017 Feb 27. PMID 28249828
- [Background] Kang J, Whang K, Hong SK, Pyen JS, Cho SM, Kim JY, Kim SH, Oh JW. Middle Meningeal Artery Embolization in Recurrent Chronic Subdural Hematoma Combined with Arachnoid Cyst. Korean J Neurotrauma. 2015 Oct;11(2):187-90. doi: 10.13004/kjnt.2015.11.2.187. Epub 2015 Oct 31. PMID 27169092
- [Background] Ishihara H, Ishihara S, Kohyama S, Yamane F, Ogawa M, Sato A, Matsutani M. Experience in endovascular treatment of recurrent chronic subdural hematoma. Interv Neuroradiol. 2007 Mar 15;13 Suppl 1(Suppl 1):141-4. doi: 10.1177/15910199070130S121. Epub 2007 Jun 27. PMID 20566092
- [Background] Hirai S, Ono J, Odaki M, Serizawa T, Nagano O. Embolization of the Middle Meningeal Artery for Refractory Chronic Subdural Haematoma. Usefulness for Patients under Anticoagulant Therapy. Interv Neuroradiol. 2004 Dec 24;10 Suppl 2(Suppl 2):101-4. doi: 10.1177/15910199040100S218. Epub 2008 May 15. PMID 20587257
- [Background] Hashimoto T, Ohashi T, Watanabe D, Koyama S, Namatame H, Izawa H, Haraoka R, Okada H, Ichimasu N, Akimoto J, Haraoka J. Usefulness of embolization of the middle meningeal artery for refractory chronic subdural hematomas. Surg Neurol Int. 2013 Aug 19;4:104. doi: 10.4103/2152-7806.116679. eCollection 2013. PMID 24032079
- [Background] Chihara H, Imamura H, Ogura T, Adachi H, Imai Y, Sakai N. Recurrence of a Refractory Chronic Subdural Hematoma after Middle Meningeal Artery Embolization That Required Craniotomy. NMC Case Rep J. 2014 May 9;1(1):1-5. doi: 10.2176/nmccrj.2013-0343. eCollection 2014 Oct. PMID 28663942
- [Background] Mauskopf JA, Sullivan SD, Annemans L, Caro J, Mullins CD, Nuijten M, Orlewska E, Watkins J, Trueman P. Principles of good practice for budget impact analysis: report of the ISPOR Task Force on good research practices--budget impact analysis. Value Health. 2007 Sep-Oct;10(5):336-47. doi: 10.1111/j.1524-4733.2007.00187.x. PMID 17888098
- [Background] Sullivan SD, Mauskopf JA, Augustovski F, Jaime Caro J, Lee KM, Minchin M, Orlewska E, Penna P, Rodriguez Barrios JM, Shau WY. Budget impact analysis-principles of good practice: report of the ISPOR 2012 Budget Impact Analysis Good Practice II Task Force. Value Health. 2014 Jan-Feb;17(1):5-14. doi: 10.1016/j.jval.2013.08.2291. Epub 2013 Dec 13. PMID 24438712
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Background] Dawkins AA, Evans AL, Wattam J, Romanowski CA, Connolly DJ, Hodgson TJ, Coley SC. Complications of cerebral angiography: a prospective analysis of 2,924 consecutive procedures. Neuroradiology. 2007 Sep;49(9):753-9. doi: 10.1007/s00234-007-0252-y. Epub 2007 Jun 27. PMID 17594083
- [Background] Fifi JT, Meyers PM, Lavine SD, Cox V, Silverberg L, Mangla S, Pile-Spellman J. Complications of modern diagnostic cerebral angiography in an academic medical center. J Vasc Interv Radiol. 2009 Apr;20(4):442-7. doi: 10.1016/j.jvir.2009.01.012. Epub 2009 Feb 26. PMID 19246211
- [Background] Kaufmann TJ, Huston J 3rd, Mandrekar JN, Schleck CD, Thielen KR, Kallmes DF. Complications of diagnostic cerebral angiography: evaluation of 19,826 consecutive patients. Radiology. 2007 Jun;243(3):812-9. doi: 10.1148/radiol.2433060536. PMID 17517935
- [Background] Link TW, Rapoport BI, Paine SM, Kamel H, Knopman J. Middle meningeal artery embolization for chronic subdural hematoma: Endovascular technique and radiographic findings. Interv Neuroradiol. 2018 Aug;24(4):455-462. doi: 10.1177/1591019918769336. Epub 2018 May 2. PMID 29720020
- See also: Efficacy of Atorvastatin in Chronic Subdural Haematoma (REACH). — https://clinicaltrials.gov/ct2/show/NCT03956368?cond=Chronic+Subdural+Hematoma&draw=2&rank=5.
- See also: Tranexamic Acid to Prevent OpeRation in Chronic Subdural Hematoma — https://clinicaltrials.gov/ct2/show/NCT03582293?cond=Chronic+Subdural+Hematoma&draw=2&rank=30.
- See also: Tocilizumab (RoActemra) and Tranexamic Acid (Cyklokapron) Used as Adjuncts to Chronic Subdural Hematoma Surgery. — https://clinicaltrials.gov/ct2/show/NCT03353259?cond=Chronic+Subdural+Hematoma&draw=2&rank=17.
- See also: Tranexamic Acid in the Treatment of Residual Chronic Subdural Hematoma (TRACE). — https://clinicaltrials.gov/ct2/show/NCT03280212?cond=Chronic+Subdural+Hematoma&draw=2&rank=4.
- See also: Treatment of Chronic Subdural Hematoma by Corticosteroids (SUCRE) — https://clinicaltrials.gov/ct2/show/NCT02650609?cond=Chronic+Subdural+Hematoma&draw=2&rank=1.
- See also: Guideline for economic evaluations in healthcare — https://english.zorginstituutnederland.nl/about-us/working-methods-and-procedures/guideline-for-economic-evaluations-in-healthcare
- See also: Code of Conduct for Medical Research — https://english.ccmo.nl/investigators/legal-framework-for-medical-scientific-research/codes-of-conduct/code-of-conduct-for-health-research